CLINICAL TRIAL: NCT05542862
Title: Immunogenicity and Safety Study in Ambulatory Adults of a Single Intramuscular Dose of SpikoGen Vaccine as a Heterologous or Homologous Booster Dose Following Completion of a Primary Course of Covid-19 Vaccine
Brief Title: Booster Study of SpikoGen COVID-19 Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Australian Respiratory and Sleep Medicine Institute Ltd (Unknown); Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AUST-C19-booster
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: covid-19; vaccine; adjuvant; Spikogen; Advax; CpG55.2
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine

STUDY DESIGN:
Intervention Model Description: All subjects will receive the same single intervention with analysis groups being based on the type of primary vaccine received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpikoGen vaccine (Experimental): Single booster dose of SpikoGen Covid-19 vaccine
  Interventions: Biological: SpikoGen vaccine

INTERVENTIONS:
Biological: SpikoGen vaccine — Recombinant spike protein based Covid-19 vaccine
  Other Names: Covax-19

SUMMARY:
The purpose of the study is to assess the effectiveness of Spikogen vaccine when used as a 3rd or 4th dose booster in adults who have been previously vaccinated with any Covid-19 vaccine types, including mRNA vaccine, adenoviral vector vaccines, recombinant protein vaccines, or inactivated virus vaccines.

DETAILED DESCRIPTION:
Currently in Australia, mRNA, adenoviral vector and recombinant protein vaccines have provisional approval for use as 3rd or 4th booster doses. This study will provide important data on the use of Spikogen as an alternative recombinant protein booster vaccine. The study will provide data in ambulatory adults on the safety and effectiveness of Spikogen vaccine when administered as a single intramuscular booster dose in those who previously vaccinated with mRNA vaccine in comparison to those immunised with other Covid-19 vaccine platforms.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Males or females 18 years of age or older
* Have previously had a primary course of Covid-19 vaccine with the most recent dose no less than 3 months previously.
* Understand and are likely to comply with planned study procedures and be available for all study visits.

Exclusion Criteria

* Allergy to Spikogen vaccine or one of its components, e.g. polysorbate 80.
* Have received an experimental agent within 30 days prior to the study vaccination or expect to receive another experimental agent during the trial reporting period.
* Any serious medical, social or mental condition which, in the opinion of the investigator, would be detrimental to the subjects or the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Seroconversion | Between baseline and 4 weeks post the booster dose
  Proportion of study participants who seroconvert (4-fold or greater rise in serum spike antibody) by primary vaccine group
Seroprotection | Between baseline and 4 weeks post the booster dose
  Proportion of study participants who achieve a spike protein neutralisation titer of 32 or greater by primary vaccine group
Geometric mean titer fold change | Between baseline and 4 weeks post the booster dose
  Increase in Geometric mean titer of spike neutralisation antibodies by primary vaccine group
Safety assessment 1 | Occurring within 7 days after booster dose.
  Frequency of Adverse events by primary vaccine group
Safety assessment 2 | Between time of administration of booster dose and through study completion, an average of 3 months
  Frequency of Serious Adverse events by primary vaccine group
SARS-CoV-2 infection | Between time of administration of booster dose and through study completion, an average of 3 months
  Frequency of SARS-CoV-2 infections in study participants by primary vaccine group, age, gender, co-morbidities, and past infection
Antibody durability | Between time of administration of booster dose and through study completion, an average of 3 months
  The proportion of subjects who remain seroprotected throughout the duration of the study including broken down by primary vaccine group.
Seroconversion in participants with and without evidence of past infection | Between baseline and 4 weeks post the booster dose and through study completion, an average of 3 months
  Spike antibody seroconversion in baseline nuclear protein antibody positive versus negative participants by primary vaccine group
Seroprotection in participants with and without evidence of past infection | Between baseline and 4 weeks post the booster dose and through study completion, an average of 3 months
  Spike antibody seroprotection in baseline nuclear protein antibody positive versus negative participants by primary vaccine group
Spike antibody GMT in participants with and without evidence of past infection | Between baseline and 4 weeks post the booster dose and through study completion, an average of 3 months
  Spike antibody GMT in baseline nuclear protein antibody positive versus negative participants by primary vaccine group.

SECONDARY OUTCOMES:
Antibody correlates of protection | Baseline and 4 weeks post the booster dose, and through study completion, an average of 3 months
  SARS-CoV-2 antibody levels in subjects with or without breakthrough SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Sajkov, MD/PhD, Principal Investigator — ARASMI; Nikolai Petrovsky, MD/PhD, Study Director — Vaxine Pty Ltd
Locations (1):
- ARASMI, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tabarsi P, Anjidani N, Shahpari R, Mardani M, Sabzvari A, Yazdani B, Roshanzamir K, Bayatani B, Taheri A, Petrovsky N, Li L, Barati S. Safety and immunogenicity of SpikoGen(R), an Advax-CpG55.2-adjuvanted SARS-CoV-2 spike protein vaccine: a phase 2 randomized placebo-controlled trial in both seropositive and seronegative populations. Clin Microbiol Infect. 2022 Sep;28(9):1263-1271. doi: 10.1016/j.cmi.2022.04.004. Epub 2022 Apr 15. PMID 35436611
- [Background] Tabarsi P, Anjidani N, Shahpari R, Roshanzamir K, Fallah N, Andre G, Petrovsky N, Barati S. Immunogenicity and safety of SpikoGen(R), an adjuvanted recombinant SARS-CoV-2 spike protein vaccine as a homologous and heterologous booster vaccination: A randomized placebo-controlled trial. Immunology. 2022 Nov;167(3):340-353. doi: 10.1111/imm.13540. Epub 2022 Jul 13. PMID 35758850
- [Background] Li L, Honda-Okubo Y, Baldwin J, Bowen R, Bielefeldt-Ohmann H, Petrovsky N. Covax-19/Spikogen(R) vaccine based on recombinant spike protein extracellular domain with Advax-CpG55.2 adjuvant provides single dose protection against SARS-CoV-2 infection in hamsters. Vaccine. 2022 May 20;40(23):3182-3192. doi: 10.1016/j.vaccine.2022.04.041. Epub 2022 Apr 18. PMID 35465982
- [Background] Li L, Honda-Okubo Y, Huang Y, Jang H, Carlock MA, Baldwin J, Piplani S, Bebin-Blackwell AG, Forgacs D, Sakamoto K, Stella A, Turville S, Chataway T, Colella A, Triccas J, Ross TM, Petrovsky N. Immunisation of ferrets and mice with recombinant SARS-CoV-2 spike protein formulated with Advax-SM adjuvant protects against COVID-19 infection. Vaccine. 2021 Sep 24;39(40):5940-5953. doi: 10.1016/j.vaccine.2021.07.087. Epub 2021 Aug 3. PMID 34420786
- [Background] Tabarsi P, Anjidani N, Shahpari R, Mardani M, Sabzvari A, Yazdani B, Kafi H, Fallah N, Ebrahimi A, Taheri A, Petrovsky N, Barati S. Evaluating the efficacy and safety of SpikoGen(R), an Advax-CpG55.2-adjuvanted severe acute respiratory syndrome coronavirus 2 spike protein vaccine: a phase 3 randomized placebo-controlled trial. Clin Microbiol Infect. 2023 Feb;29(2):215-220. doi: 10.1016/j.cmi.2022.09.001. Epub 2022 Sep 10. PMID 36096430
- [Derived] Honda-Okubo Y, Sajkov D, Wauchope B, Turner JV, Vote B, Antipov A, Andre G, Lebedin Y, Petrovsky N. Immunogenicity and safety study of a single dose of SpikoGen(R) vaccine as a heterologous or homologous intramuscular booster following a primary course of mRNA, adenoviral vector or recombinant protein COVID-19 vaccine in ambulatory adults. Vaccine. 2025 Mar 7;49:126744. doi: 10.1016/j.vaccine.2025.126744. Epub 2025 Feb 5. PMID 39914274